CLINICAL TRIAL: NCT02657629
Title: Comparison of Feeding Strategies After Stage 1 Procedures for Hypoplastic Left Heart Syndrome Infants: A Randomized Controlled Trial
Brief Title: Comparison of Feeding Strategies for Hypoplastic Left Heart Syndrome Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Nicole Spillane, Pediatric Fellow, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAE0781
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Hypoplastic Left Heart Syndrome; Growth Failure
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Failure to Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Feeding Regimen (Active Comparator): Enteral feedings given as combination of continuous nocturnal feedings and intermittent bolus daytime feedings.
  Interventions: Other: Continuous Feeding Regimen
- Intermittent Bolus Feeding Regimen (Active Comparator): Enteral feedings given as intermittent bolus feedings for entire 24 hour period.
  Interventions: Other: Intermittent Bolus Feeding Regimen

INTERVENTIONS:
Other: Continuous Feeding Regimen — Nocturnal continuous enteral feedings given from 8pm-8am with intermittent bolus feedings every 3 hours between 11am and 5pm. Continuous feedings given via gavage (nasogastric tube, orogastric tube or gastrostomy tube) and intermittent bolus feeds via gavage or nipple. Total caloric intake maintained at 120-130 kcal/kg/d.
  Arms: Continuous Feeding Regimen
Other: Intermittent Bolus Feeding Regimen — Intermittent bolus enteral feedings given after 3 hours for entire 24 hours period. Feedings given via gavage or nipple. Total caloric intake maintained at 120-130 kcal/kg/d.
  Arms: Intermittent Bolus Feeding Regimen

SUMMARY:
The purpose of the study is to determine if a continuous feeding regimen as compared to an intermittent bolus feeding regimen leads to improved weight gain in infants with hypoplastic left heart syndrome (HLHS) after stage 1 procedures.

DETAILED DESCRIPTION:
In recent years, survival after neonatal cardiac surgery has improved significantly. As life span has improved in HLHS/single ventricle variants (SVV) survivors, focus has shifted to the understanding and management of associated health problems. Growth failure is a well-recognized major co-morbidity in these patients.

Infants with HLHS/SVV demonstrate progressive growth failure after stage 1 procedures, which appears to stabilize only after stage 2 procedures. Poor nutritional status increases risk for post-operative infections, extends hospital length-of-stay, and adversely affects neurodevelopmental outcomes.

To date, evidence-based feeding strategies that support adequate weight gain and improve nutritional status have not been identified after stage 1 procedures. Continuous enteral feeding regimens have resulted in improved growth in a diverse population of infants with congenital heart disease and have been shown to decrease energy expenditure in premature infants and adults. A randomized, controlled study of HLHS/SVV infants who underwent stage 1 procedures at a single medical center was conducted with the primary objective of comparing weight gain at hospital discharge between infants receiving a continuous feeding regimen versus an intermittent feeding regimen. Secondary objectives were to compare growth and markers of nutritional status at hospital discharge between the two groups. The investigators hypothesized that infants with HLHS/SVV who receive a continuous enteral feeding regimen versus an intermittent feeding regimen will demonstrate improved weight gain, growth, and nutritional status after stage 1 procedures at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with HLHS/SVV who underwent stage 1 procedures (Norwood or Hybrid procedure) who were inborn or transferred into the Neonatal Intensive Care Unit at Columbia University Medical Center

Exclusion Criteria:

- Excluded subjects were those with associated major congenital malformations (e.g. congenital diaphragmatic hernia, gastroschisis) or chromosomal anomalies, and/or those who were small for gestational age at birth.

- Subjects in whom a nasogastric tube or gastrostomy tube was not required for feeding at the time of enrollment and/or who were transferred to outside institutions for recovery after surgery.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2009-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ganga Krishnamurthy, MD, Principal Investigator — Columbia University

REFERENCES:
- [Background] Slicker J, Hehir DA, Horsley M, Monczka J, Stern KW, Roman B, Ocampo EC, Flanagan L, Keenan E, Lambert LM, Davis D, Lamonica M, Rollison N, Heydarian H, Anderson JB; Feeding Work Group of the National Pediatric Cardiology Quality Improvement Collaborative. Nutrition algorithms for infants with hypoplastic left heart syndrome; birth through the first interstage period. Congenit Heart Dis. 2013 Mar-Apr;8(2):89-102. doi: 10.1111/j.1747-0803.2012.00705.x. Epub 2012 Aug 14. PMID 22891735
- [Result] Wolovits JS, Torzone A. Feeding and nutritional challenges in infants with single ventricle physiology. Curr Opin Pediatr. 2012 Jun;24(3):295-300. doi: 10.1097/MOP.0b013e32835356ae. PMID 22572758
- [Result] Grant J, Denne SC. Effect of intermittent versus continuous enteral feeding on energy expenditure in premature infants. J Pediatr. 1991 Jun;118(6):928-32. doi: 10.1016/s0022-3476(05)82213-9. PMID 1904091
- [Result] Heymsfield SB, Casper K, Grossman GD. Bioenergetic and metabolic response to continuous v intermittent nasoenteric feeding. Metabolism. 1987 Jun;36(6):570-5. doi: 10.1016/0026-0495(87)90169-7. PMID 3108622
- [Result] Ravishankar C, Zak V, Williams IA, Bellinger DC, Gaynor JW, Ghanayem NS, Krawczeski CD, Licht DJ, Mahony L, Newburger JW, Pemberton VL, Williams RV, Sananes R, Cook AL, Atz T, Khaikin S, Hsu DT; Pediatric Heart Network Investigators. Association of impaired linear growth and worse neurodevelopmental outcome in infants with single ventricle physiology: a report from the pediatric heart network infant single ventricle trial. J Pediatr. 2013 Feb;162(2):250-6.e2. doi: 10.1016/j.jpeds.2012.07.048. Epub 2012 Aug 30. PMID 22939929
- [Result] Hehir DA, Cooper DS, Walters EM, Ghanayem NS. Feeding, growth, nutrition, and optimal interstage surveillance for infants with hypoplastic left heart syndrome. Cardiol Young. 2011 Dec;21 Suppl 2:59-64. doi: 10.1017/S1047951111001600. PMID 22152530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Feeding Regimen | Intermittent Bolus Feeding Regimen
Started | 14 | 14
Completed | 12 | 14
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Feeding Regimen | Intermittent Bolus Feeding Regimen | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 14 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: gestational age in weeks at birth] | 38.3 (1) | 38.9 (1.5) | 38.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain in Grams Per Day
Time Frame: Daily until hospital discharge (up to maximum of 3 months of age)
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Continuous Feeding Regimen | Intermittent Bolus Feeding Regimen
Number analyzed (Participants) | 12 | 14
grams/day | 24.3 (14.6) | 23.6 (7.7)
Statistical Analysis 1: Comparison: Continuous Feeding Regimen vs Intermittent Bolus Feeding Regimen; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Continuous Feeding Regimen | Intermittent Bolus Feeding Regimen
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Feeding Regimen (N=12) | Intermittent Bolus Feeding Regimen (N=14)
necrotizing enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No